CLINICAL TRIAL: NCT04951362
Title: Studying the Expected Effect of Ivermectin Nanosuspension as Nasal Spray Upon Post covid19 Persistant Anosmia
Brief Title: Role of Ivermectin Nanosuspension as Nasal Spray in Treatment of Persistant Post covid19 Anosmia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Zaky Aref, ass.professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU MED CIT0 23 4 21 1 122
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intranasal Ivermectin group (Active Comparator): 49 pateints with anosmia received ivermectin nanosuspension nasal spray
  Interventions: Drug: intranasal spray ivermectin
- saline nasal spray (Placebo Comparator): 47 pateints with anosmia received saline nasal spray
  Interventions: Drug: intranasal spray ivermectin

INTERVENTIONS:
Drug: intranasal spray ivermectin — intranasal spray of saline
  Other Names: saline spray

SUMMARY:
ivermectin is FDA approaved antiparasitic drug which is also claimed to be having potent in vitro antiviral effect,so we are tryying to study itsovid19 anosmia effect upon releiving post covid19 anosmia

DETAILED DESCRIPTION:
ivermectin is FDA approaved antiparasitic drug which is also claimed to be having potent in vitro antiviral effect,so we are tryying to study itsovid19 anosmia effect upon releiving post covid19 anosmia as one of the most characteresic symptoms of covid19 infection

ELIGIBILITY:
Inclusion Criteria:

* post covid19 anosmia
* negative swab test for covid19

Exclusion Criteria:

* other types of anosmia ,
* no local or central other causes of anosmia
* still active covid 19 pateints ( positive swab test )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-05-12 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
regaining of smell | within 14 days after enrollemen ]
  regaining of smell

CONTACTS AND LOCATIONS:
Locations (1):
- Zaky Aref, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aref ZF, Bazeed SEES, Hassan MH, Hassan AS, Ghweil AA, Sayed MAA, Rashad A, Mansour H, Abdelmaksoud AA. Possible Role of Ivermectin Mucoadhesive Nanosuspension Nasal Spray in Recovery of Post-COVID-19 Anosmia. Infect Drug Resist. 2022 Sep 19;15:5483-5494. doi: 10.2147/IDR.S381715. eCollection 2022. PMID 36164334